CLINICAL TRIAL: NCT05475171
Title: Triage of Advanced Cervical Cancer Through Immunotherapy Induction (TRACTION)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0107; NCI-2022-06116 (Other: NCI-CTRP Clinical Trias)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Cancer; Cervical Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lorigerlimab (Experimental): Participants will receive Lorigerlimab by vein over about 30 minutes on Day 1 of each cycle
  Interventions: Drug: Lorigerlimab

INTERVENTIONS:
Drug: Lorigerlimab — Given by vein (IV)
  Other Names: MGD019

SUMMARY:
To learn if MGD019 can help to control cervical cancer in patients who have yet to receive treatment.

DETAILED DESCRIPTION:
Primary Objectives:

To estimate disease control rate (DCR) in patients with metastatic, recurrent, or persistent cervical cancer who have not received prior systemic chemotherapy and are undergoing induction immunotherapy with MGD019.

Secondary Objectives:

1. To determine overall survival (OS)
2. To determine progression-free survival (PFS)
3. To determine objective response rate (ORR)
4. To determine duration of response (DOR)
5. To evaluate safety of administering MGD019 in cervical cancer patients using the National Institute of Health Common Terminology Criteria for Adverse Events (CTCAE) v5.0

Exploratory Objectives:

1. To investigate molecular and immunological changes in the tumor tissue prior to and on-treatment with MGD019
2. To identify treatment-induced tissue-based alterations in malignant and immune cells and their correlation with response, progression, and immune-related adverse events
3. To determine the utility of cell-free DNA for evaluation treatment response

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be assessed within 28 days of starting study treatment:

1. Ability to provide signed informed consent
2. Age ≥ 18 years at time of study entry
3. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
4. Biopsy or CT scan confirmed recurrent, metastatic, or persistent cervical cancer
5. One of the following histologic subtypes: squamous cell carcinoma, adenosquamous, or adenocarcinoma
6. Not amenable to curative treatment (e.g. surgery and/or radiation)
7. Eastern Cooperative Oncology Group performance status 0 - 1
8. Measurable disease by RECIST v1.1
9. Adequate normal organ and marrow function as defined below.

   1. Hemoglobin ≥8.0 g/dL.
   2. Absolute neutrophil count (ANC) > 1000/mm3

      .
   3. Platelet count ≥100 x 109

      /L (>75,000/mm3

      ).
   4. Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   5. AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN.
   6. International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
   7. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiationinduced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. If vaccinated against COVID-19, the last vaccine dose must be 14 days or greater from the first investigational product administration.
12. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the PI

Exclusion Criteria:

Exclusion criteria will be assessed within 28 days of starting study treatment:

1. Prior systemic chemotherapy except when used with concurrent radiation therapy
2. Is pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
3. Previous immune checkpoint inhibitor therapy or cytokines
4. Ongoing or active systemic infection, active hepatitis B or C infection, or known uncontrolled HIV, that might affect host immunity. Patients with stable, controlled HIV (defined as CD4+ T-cell counts ≥ 350 cells/uL, on established antiretroviral therapy for at least 4 weeks, and have an HIV viral load less than 400 copies/mL prior to enrollment) are eligible for trial inclusion.
5. History of chronic obstructive pulmonary disease or other intrinsic lung disease requiring systemic steroid therapy, oxygen, or hospitalization
6. History of clinically significant cardiovascular disease or QTcF > 470 within 12 months from first dose of study intervention, including New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular event, or cardiac arrhythmia associated with hemodynamic instability. Note: medically controlled arrhythmia would be permitted.
7. History of immunodeficiency or receiving chronic systemic steroid or other immunosuppressive therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Steroid premedications for radiologic contrast allergy are permitted.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Has history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
11. Other illnesses/conditions that in the investigator's opinion would adversely affect the safety of checkpoint inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To establish overall survival (OS) | through the study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazeri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org